CLINICAL TRIAL: NCT02620826
Title: Prospective Comparison of Indirect Pulp Therapy and Mineral Trioxide Aggregate Pulpotomy in Decayed Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James R. Boynton, Clinical Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00077025
Record Dates: First submitted 2015-01-28; First posted 2015-12-03 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dental Pulp Capping
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indirect pulp therapy (Experimental): Primary molars will be treated with indirect pulp therapy using resin-modified glass ionomer (Vitrebond Plus).
  Interventions: Procedure: Indirect pulp therapy
- Pulpotomy (Active Comparator): Primary molars treated with MTA pulpotomy.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Indirect pulp therapy — Decayed dentin is lined with a resin-modified glass ionomer (Vitrebond Plus)
  Arms: Indirect pulp therapy
Procedure: Pulpotomy — A cervical pulpotomy is done and the radicular pulp is lined with Mineral Trioxide Aggregate
  Arms: Pulpotomy

SUMMARY:
This prospective study compares the use of indirect pulp therapy and mineral trioxide aggregate pulpotomy for pulp therapy of the primary molar with dental caries approaching the pulp.

ELIGIBILITY:
Inclusion Criteria:

* Child with at least one primary molar with deep decay approaching the pulp.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2013-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Clinical assessment of pulp vitality | 10 years
  Pain, mobility, abscess as determined with clinical evaluation

SECONDARY OUTCOMES:
Radiographic assessment of pulp vitality | 10 years
  Signs of pulpal degeneration, including evaluation for presence or absence of internal/external root resorption, periodontal ligament widening, and intraradicular radiolucency as determined with radiographic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States